CLINICAL TRIAL: NCT02735330
Title: Intra Operative Coeliac Plexus Neurolysis Combined With Frey's Procedure for Effective Pain Relief in Patients With Chronic Calcific Pancreatitis- A Prospective Randomized Double-blind Placebo Controlled Trial
Brief Title: Intraoperative Coeliac Plexus Alcohol Neurolysis Along With Frey's Procedure for a Better Pain Relief
Acronym: INFARCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Madras Medical College (Other Government)
Responsible Party: Principal Investigator, Balakumaran Sathyamoorthy, Principal investigator, Madras Medical College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ID-NO 23052015; CTRI/2016/02/006593 (Registry Identifier: Clinical trial registry India.)
Record Dates: First submitted 2016-03-16; First posted 2016-04-12 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Calcific Pancreatitis
Keywords: CCP
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GROUP 1 (Active Comparator): 68 Patients undergo Frey's procedure with celiac plexus neurolysis using absolute alcohol
  Interventions: Procedure: celiac plexus neurolysis using absolute alcohol; Procedure: Frey's procedure
- GROUP 2 (Placebo Comparator): 68 Patients undergo Frey's procedure with Placebo celiac plexus injection using saline
  Interventions: Procedure: Placebo celiac plexus injection using saline; Procedure: Frey's procedure

INTERVENTIONS:
Procedure: celiac plexus neurolysis using absolute alcohol — celiac plexus blockade with 40 ml of diluted absolute alcohol(50%) 20 ml on either side of celiac axis in a 4 quadrant fashion
  Other Names: NCPB, Neurolytic celiac plexus block
  Arms: GROUP 1
Procedure: Placebo celiac plexus injection using saline — Placebo celiac plexus injection with 40 ml of saline 20 ml on either side of celiac axis in a 4 quadrant fashion for blinding
  Other Names: Placebo
  Arms: GROUP 2
Procedure: Frey's procedure — Pancreatic head is partially resected (cored) along with longitudinal opening of duct along its entire length with limit of excavation of the head in the plane of the posterior wall of the Wirsung's duct and duct of Santorini is opened in the uncinate process. All the tissue above the plane, including the duct of Santorini is excised. The reconstruction is done with covering with a loop of jejunum in Roux-en-Y fashion which continues with the main pancreatic duct in the pancreatic body and tail.
  Other Names: Duodenum preserving pancreatic head coring procedure

SUMMARY:
To study the effect of Intra operative Coeliac plexus alcohol neurolysis combined with Frey's procedure for effective pain relief in patients with Chronic Calcific Pancreatitis in a single centre setting with a Randomized Controlled Trial.

DETAILED DESCRIPTION:
165 consecutive CCP patients admitted in our surgical gastro enterology department since January 2013 were screened for eligibility. 29 patients were excluded (28 were not meeting the inclusion criteria and 1 patient intra operatively found to have disseminated malignancy). After exclusion 136 patients were included in our study. They were randomized in to 2 groups, one group was treated by Frey's procedure with NCPB (Group-I) and the other by Frey's procedure with saline as placebo (Group-II). Method of Study is a randomized, double- blind, placebo- controlled, parallel arm, superiority trial.

Randomization was done at the time of surgery using random number table created with computerized software by a statistician not involved in this study.

Blinding and masking was done by using pre numbered containers having filled with either absolute alcohol or saline according to the randomization chart which was then kept sealed by an office staff until the end of the study. Both subjects and response assessor were blinded.

Data collection:

The preoperative baseline details such as etiology, morphology, associated complications and VAS pain score, Izbicki pain score, weight loss, insulin requirement, LFT (liver function tests), serum amylase & lipase, fasting sugar& fecal elastase were collected on admission.

Additional procedures, presence of peripancreatic inflammatory changes (fibrosis) as evidenced by difficult Kocherisation and plasted capsule and intra-operative complications were noted during surgery.

Short term follow up details including pain relief measured by VAS score &Izbicki pain score, analgesic consumption, weight gain, improvement in steatorrhoea (Fecal elastase>200 µg/g of stool & subjective reduction in foul smelling oily diarrhea), diabetic status (fasting glucose, GTT, HgbA1c, insulin& oral hypoglycemic agents requirement), mortality and morbidity were noted.

Follow up details were collected every 3 months as outpatient basis. Standard questionnaire format of SF 12 Version-2 was used for QOL assessment every 6 months in a face to face interview.

Statistical analysis was performed in SPSS version 20. Continuous variables were presented as mean, standard deviation and 95% confidence interval; categorical variables were presented as frequencies. The chi-square test and the Fisher exact test were used to analyze categorical variables. The unpaired Student t test was used to analyze continuous variables. P value <0.05 was considered statistically significant. Factors found significant on univariate logistic regression analysis were incorporated in to the multivariate logistic regression analysis for odds ratio with 95% confidence intervals to analyze the significant factors affecting the outcome of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive chronic calcific pancreatitis admitted in our institute since 2013 january with age group between 13 to 65 years with Visual analogue scale (VAS) pain score of more than 7 and those who have quit alcohol & smoking for at least 6 months are included in our study.

Exclusion Criteria:

* Patients with mild to moderate pain score (VAS pain score 1-7), continuous substance abuse, severe comorbid illness are excluded from study.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Pain relief measured by Visual Analogue Scale | up to 5 years
  Short term (2 years) and long term(5 years) score at follow up at out patient clinic or over phone.

SECONDARY OUTCOMES:
Number of patients with improvement in endocrine function as measured by Fasting glucose of < 130 and HbA1c level of <6.5% | up to 5 years
  and reduction in dosage of insulin (iu) & oral hypoglycemic agents (milli gm) when compared to preoperative levels- at out patient clinic
Number of patients with improvement or worsening in exocrine function as measured by the estimation of fecal elastase >200 µg/g of stool or <200 µg/g of stool respectively at out patient clinic. | up to 5 years
Analgesics intake | up to 5 years
  Dosage and frequency of intake of both NSAIDs and opioid analgesics intake are noted at out patient clinic or over phone.
Weight gain in kg measured at out patient clinic | up to 5 years
Quality of life | up to 5 years
  Using SF 12 V2 (Tamil and english version-Optuminsight Life Sciences) in a face to face (written form) interview at out patient clinic
Number of patients with worsening in endocrine function as measured by abnormal laboratory values like Fasting glucose >130 and HbA1c >6.5 | up to 5 years
  and increased dosage of insulin (IU)& oral hypoglycemic agents(milli gms) requirement when compared to preoperative levels at out patient clinic
Number of patients with abnormal lab values like Fasting glucose of >126 mg/dl or blood glucose level of >200 after a standard glucose tolerance test (GTT) in equivocal cases. | up to 5 years

OTHER OUTCOMES:
Frequency of pain attacks | Up to 5 years
  whether pain attacks are occurring in a daily/several times in a week/month/Year is noted.
Time of disease related inability to work | Up to 5 years
  Whether the restriction of work activities last permanently/ Up to 1 year/month/week or no restriction is noted
Type of analgesic medication (morphine related analgesic potency) | Up to 5 years
  What analgesic medication is taken by the patient like morphine,pethidine,buprenorphine, tramadol,aspirin, paracetamol are noted.

CONTACTS AND LOCATIONS:
Overall Officials: KANNAN DEVYGOUNDER, MS,MCh,FRCS, Study Director — MADRAS MEDICAL COLLEGE,CHENNAI,TAMIL NADU,INDIA; BALAKUMARAN SATHYAMOORTHY, Principal Investigator — MADRAS MEDICAL COLLEGE,CHENNAI,TAMIL NADU, INDIA

IPD SHARING:
Plan to Share IPD: Yes
with out showing the name of the participants we can disclose the data of the all participants